CLINICAL TRIAL: NCT06068517
Title: Closed Incision Negative Pressure Wound Therapy for the Prevention of Surgical Site Infections in Abdominal Surgery - A Multicenter Randomized Controlled Trial
Brief Title: Closed Incision Negative Pressure Wound Therapy for the Prevention of Surgical Site Infections in Abdominal Surgery
Acronym: CISSI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Clinical Trials Unit University of Bern (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CISSI
Record Dates: First submitted 2023-09-27; First posted 2023-10-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Surgical Wound Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed incision negative pressure wound therapy (Experimental): At the completion of the surgical procedure, the skin will be closed with staples at a distance of two centimeters from each other. After skin closure, ciNPWT will be applied, using a commercially available device. The device will be left in place for 7 days.
  Interventions: Device: Closed incision negative pressure wound therapy
- Standard dressing (Active Comparator): At the completion of the surgical procedure, the skin will be closed with staples at a distance of two centimeters from each other. After skin closure, conventional dry dressings will be applied. Conventional dressings will be changed according to clinical practice in the participating study centers.
  Interventions: Device: Standard dressing

INTERVENTIONS:
Device: Closed incision negative pressure wound therapy — After the completion of abdominal surgery and standardised skin closure with staples, ciNPWT will be applied, using a commercially available device.
  Arms: Closed incision negative pressure wound therapy
Device: Standard dressing — After the completion of abdominal surgery and standardised skin closure with staples, standard dressings will be applied.
  Arms: Standard dressing

SUMMARY:
Surgical site infections (SSI) are a frequent complication in abdominal surgery. SSI lead to worse outcomes for the affected patients and significantly higher healthcare costs. Closed incision negative pressure wound therapy (ciNPWT) consists of a non-invasive, vacuum-assisted system that applies negative pressure to closed surgical incisions. It is currently unclear, if ciNPWT reduces SSI in patients undergoing abdominal surgery. This trial will investigate the effect of ciNPWT on SSI in abdominal surgery.

DETAILED DESCRIPTION:
Background:

Surgical site infections (SSI) are a frequent complication after abdominal surgery and are associated with increased morbidity and mortality, longer hospital stay, and significantly increased healthcare costs. Closed incision negative pressure wound therapy (ciNPWT) is a non-invasive, vacuum-assisted system that applies negative pressure to closed surgical incisions. Recent meta-analyses suggest that ciNPWT reduces the risk of SSI in abdominal surgery. However, based on the available randomized controlled trials (RCT), the evidence for the effect of ciNPWT on SSI in abdominal surgery is insufficient.

Rationale:

Considering the frequent occurrence of SSI in abdominal surgery, associated worse outcomes, and insufficient evidence, an adequately powered, robust RCT investigating the effect of ciNPWT on SSI in elective and emergency abdominal surgery is warranted. Provided that ciNPWT significantly reduces the incidence of SSI, this adjunct to surgical therapy has the potential to fundamentally improve patient outcomes in abdominal surgery.

Aim of the trial:

To investigate the effect of ciNPWT on superficial and deep SSI in patients undergoing elective or emergency abdominal surgery by laparotomy.

Methodology:

Multicenter, open-label, two arm, parallel group RCT. Patients undergoing elective or emergency laparotomy will be enrolled. During surgery, participants will be randomized in a 1:1 ratio to the ciNPWT (treatment) or standard dressing (control) group. After the completion of abdominal surgery and standardized skin closure with staples, either ciNPWT or standard dry dressings will be applied. Other than the study procedure, participants in both groups will be treated the same according to the current standard of care at the participating centers. Data collection will be carried out during the subsequent hospital stay and at 30 (+/- 7) days postoperatively.

Hypothesis:

The investigators hypothesize that ciNPWT will significantly reduce the incidence of superficial and deep SSI in patients undergoing laparotomy.

ELIGIBILITY:
Inclusion Criteria:

* Elective or emergency laparotomy, or laparoscopy converted to laparotomy, including surgery for complications after elective operations
* Incision length ≥ 10 cm
* Centers for Disease Control and Prevention (CDC) wound class 1 and 2 (clean, clean-contaminated)
* Abdominal closure with or without mesh implantation
* Primary abdominal closure or closure after open abdomen treatment
* Age over 18 years
* Written informed consent

Exclusion Criteria:

* Age ≤ 18 years
* CDC wound class 4 (dirty/infected wound)
* Organ transplantation
* Sensitivity or allergy to silver

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 654 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Composite incidence of superficial and deep surgical site infections | 30 (+/- 7) days
  Number of participants with a superficial or deep surgical site infections at 30 (+/- 7) days postoperatively.

SECONDARY OUTCOMES:
Overall surgical site infections (superficial, deep, and organ space) | 30 (+/- 7) days
  Number of participants with a superficial or deep or organ space surgical site infections at 30 (+/- 7) days postoperatively.
Superficial, deep, and organ space surgical site infections as separate outcomes | 30 (+/- 7) days
  Number of participants with a superficial surgical site infections at 30 (+/- 7) days postoperatively.
  Number of participants with a deep surgical site infections at 30 (+/- 7) days postoperatively.
  Number of participants with an organ space surgical site infections at 30 (+/- 7) days postoperatively.
Other wound complications (wound dehiscence, seroma, hematoma) | 30 (+/- 7) days
  Number of participants with another wound complication at 30 (+/- 7) days postoperatively.
Postoperative hospital length of stay | Usually between 1 and 14 days
Duration of closed incision negative pressure wound therapy | 7 days
Number of outpatient visits | 30 days
Postoperative health-related quality of life (SF-36 Health Survey) | 30 (+/- 7) days
  Range from 0 (worst) to 100 (best).
Costs for inpatient treatment | Usually between 1 and 14 days
In-hospital mortality | Usually between 1 and 14 days
30-day mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Haltmeier, MD, Principal Investigator — Inselspital, Bern University Hospital
Locations (1):
- Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No